CLINICAL TRIAL: NCT03366493
Title: The Study of Folate Receptor-Mediated Staining Solution (FRD™) In Cervical
Brief Title: The Study of Folate Receptor-Mediated Staining Solution (FRD™) In Cervical Lesion Detection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GY Highland Biotech LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: GYFRD-001
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3
MeSH Terms: interventions — Cytological Techniques; Papanicolaou Test; Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FRD, Cyctology, HPV testing (Experimental): Subjects will be asked to have the FRD, Cytology, and HPV test performed on them by the study doctor or staff.
  Interventions: Combination Product: FRD; Other: Cytology; Other: HPV testing
- Colposcopy Examination (and ECC if necessary) (Experimental): Subjects with abnormal cytology (≥ ASCUS/AGC), positive FRD test in either the cervix or cervical canal, and/or positive HPV test will be referred to colposcopy. Subjects with a positive FRD test for the cervical canal, unsatisfied colposcopy (type II-III), and/or detection of AGC during cytology will also have to complete an ECC procedure. In addition, 10% of the subjects who tested negative for all three tests and are ≥ 25 years old will be randomly selected to complete a colposcopy as well.
  Interventions: Procedure: Colposcopy; Procedure: ECC
- Biospy (Experimental): According to the colposcopy assessment, if the results show satisfied (type I) then a biopsy will be taken. Finally, a histopathological examination will be done and used as the gold standard. Subjects with a histopathological examination result of < CIN2 will be asked to come back for a follow up visit within 6 months or 1 year, according to the investigator's discretion.
  Interventions: Procedure: Biospy

INTERVENTIONS:
Combination Product: FRD — The Folate Receptor-Mediated Staining Solution is a dye solution that stains for medical purposes used in staining cells and tissues for detecting neoplastic diseases. After inserting a speculum into your vagina, the FRD™ staining solution will be applied to the cervix using an applicator. After removal of the applicator, the doctor will inspect the applicator for color changes and note any changes. The physician will then remove any excess stain from the cervix using distilled water.
  Other Names: Folate Receptor - Mediated Staining Solution
  Arms: FRD, Cyctology, HPV testing
Other: Cytology — Cytology testing done by collecting samples of cells, and smearing those samples across a glass microscope slide in order to detect abnormal cells that may develop into cervical cancer.
  Other Names: Pap smear
  Arms: FRD, Cyctology, HPV testing
Other: HPV testing — HPV tests will detect HPV infections, which can lead to cervical cells to become cancer cells.
  Arms: FRD, Cyctology, HPV testing
Procedure: Colposcopy — During the colposcopic examination, the physician will insert a speculum into the vagina and then apply a vinegar solution to the cervix. The vinegar solution causes any potential abnormal cells to turn white. These white regions are best seen using the colposcope, which magnifiesthe skin.
  Arms: Colposcopy Examination (and ECC if necessary)
Procedure: ECC — If the examination is not satisfactory and the doctor is not able to see the entire cervix, he may perform an endocervical curettage, or ECC. This sample is collected by placing a long, thin instrument into the cervical canal and a sample is scraped from that area. The sample will be sent to the laboratory for a pathologist to review.
  Other Names: Endocervical curettage
  Arms: Colposcopy Examination (and ECC if necessary)
Procedure: Biospy — According to the colposcopy assessment, if the doctor sees a white area, or an area of abnormal cells, a tiny sample of tissue, called a biopsy will be taken from the cervix. About half of women do not feel the biopsy being taken.
  Others may feel a quick pinch. After the biopsy, the wound will be treated to stop bleeding.The biopsy will be sent to the laboratory for a pathologist to review.
  Arms: Biospy

SUMMARY:
The FRDTM is easy to perform and does not require sophisticated laboratory technology and/or experienced pathologists for test result interpretation. Compared to the Pap smear and HPV test, the FRDTM enables clinicians to obtain test results immediately (within 60 seconds) after the screening. This empowers clinicians in making timely decisions on appropriate patient management, and facilitating patient compliance with follow-up procedures. In addition, the FRDTM requires minimal training and technical support. Due to its advantage of rapid visualization of abnormal cervical lesions (CIN2+) in a cost-effective way, health care professionals can make cervical cancer detection accessible to women worldwide, especially in regions with limited medical resources. This is a cross-sectional study to evaluate the clinical performance of Folate Receptor-Mediated Epithelium Staining (FRDTM) in detecting cervical neoplastic lesions (CIN2+).

DETAILED DESCRIPTION:
The Folate Receptor-Mediated Staining Solution is a dye solution that stains for medical purposes used in staining cells and tissues for detecting neoplastic diseases. The main purpose of this product is to detect abnormal cervical lesions (CIN2+) during a gynecological speculum examination. Therefore, the purpose of this study is to evaluate the clinical performance of Folate Receptor-Mediated Epithelium Staining (FRDTM) in detecting cervical neoplastic lesions (CIN2+).

The subjects who are enrolled in this study will first undergo the FRD test, then cytology and HPV test. Women with abnormal cytology (≥ ASCUS/AGC), positive FRD test in either the cervix or cervical canal, and/or positive HPV test will be referred to colposcopy. In addition, 10% of the subjects who tested negative for all three tests and are ≥ 25 years old will be randomly selected to complete a colposcopy as well.

According to the colposcopy assessment, if the results show satisfied (type I) then a biopsy will be taken. Subjects with a positive FRD test for the cervical canal, unsatisfied colposcopy (type II-III), and/or detection of AGC during cytology will have to complete an ECC procedure as well. Finally, a histopathological examination will be done and used as the gold standard. Subjects with a histopathological examination result of < CIN2 will be asked to come back for a follow up visit within 6 months or 1 year, according to the investigator's discretion. Subjects can exit the study at any time after colposcopy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients who need to do gynecological pelvic examination
* Age and sex: Women between the ages of 20 - 65

Exclusion Criteria:

* Women with total hysterectomy
* Women who have done cervical surgeries, including physiotherapy of conization, LEEP, infrared ray, and microarray
* Women with serious cervical contact bleeding
* Women who are pregnant or menstrual period before the examination
* Women with acute inflammation of cervix and/or vagina
* Women who were already diagnosed with CIN2+
* Women who are taking an oral and/or injection of anti-cancer drugs

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Non-pregnant women who are sexually active and need to do a routine cervical cancer screening.
Enrollment: 200 (Estimated)
Dates: Start 2017-12-07 (Estimated); Primary Completion 2018-12-07 (Estimated); Study Completion 2018-12-07 (Estimated)

PRIMARY OUTCOMES:
Subjects diagnosed with CIN2+ | 2-4 weeks
  The primary outcome measure of the study is when the subjects' histological diagnosis is CIN2+. At that point they can exit the study.

SECONDARY OUTCOMES:
Subjects without CIN2+ after colposcopy | 6 months - 1 year
  The secondary outcome measures are all women < 25 years & women ≥25 years that were not chosen to be a part of the 10% with normal cytology, negative FRD, & negative HPV. Women without CIN2+ after colposcopy will have to come back for a follow up visit in 6 months or 1 year. All patients can exit the study after colposcopy.

CONTACTS AND LOCATIONS:
Overall Officials: Daron G Ferris, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided